CLINICAL TRIAL: NCT04135651
Title: Effect of Paratracheal Esophagus Pressure on the Endotracheal Intubation With Pentax Airway Scope
Brief Title: Paratracheal Esophagus Pressure on the Intubation With Pentax Airway Scope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MED-INT-19-340
Record Dates: First submitted 2019-10-15; First posted 2019-10-22 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Anesthesia; Intubation; Difficult or Failed; Cricoid Pressure; Pulmonary Aspiration During Anesthetic Induction
Keywords: Paratracheal pressure; Glottic view; Cricoid pressure; Pentax

STUDY DESIGN:
Intervention Model Description: Randomized double blinded clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The group assignments were sealed in opaque envelopes by a research assistant not involved in the study.
  The interventional process covers opaque clothes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paralaryngeal pressure (Experimental): During the induction of anesthesia, left paratracheal pressure is applied by 30N force with thumb after confirmation of the location of the esophagus using ultrasound.
  Interventions: Procedure: Paratracheal pressure
- Cricoid pressure (Active Comparator): During the induction of anesthesia, cricoid pressure is applied by 30N force with three fingers.
  Interventions: Procedure: Cricoid pressure

INTERVENTIONS:
Procedure: Paratracheal pressure — To apply paratracheal pressure, the thumb was placed over the left side of the trachea cephalad to the clavicle and medial to the sternocleidomastoid muscle.
  Arms: Paralaryngeal pressure
Procedure: Cricoid pressure — To apply cricoid pressure, the crocoid cartilage was compressed with a single-handed three-finger maneuvre towards the vertebral bodies.
  Arms: Cricoid pressure

SUMMARY:
Recently, left paratracheal pressure was introduced as an alternative method to prevent pulmonary aspiration instead of cricoid pressure. Criocoid pressure is known to worsen glottic visibility when using Pentax.However, the effects of left paratracheal pressure on glottic view when using Pentax are not studied yet. In this study, the subjects are divided into two groups (group I: left paratracheal pressure applied before intubation, group II: conventional cricoid pressure applied before intubation). Investigators will assess the glottic view during intubation using Pentax.

DETAILED DESCRIPTION:
Primary outcome

- Duration of intubation

Secondary outcomes

* POGO (percentage of glottic opening) score before and after application of each intervention
* Glottic grade by Cormack Lehane
* The success rate in first attempt
* Intubation difficulty scale
* Hemodynamics during intubation
* Postoperative airway complications

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing surgery under general anesthesia
* American Society of Anesthesiologists Classification 1-2

Exclusion Criteria:

* Body mass index > 35 kg/m2
* High risk of regurgitation (hiatus hernia, gastro-esophageal reflux disease, non-fasting status)
* Criteria for difficult airway (limitation of mouth opening/neck extension, Mallampati class IV),

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Time to intubation | During anesthesia induction procedure
  The duration from when Pentax pass the tooth to confirm the successful intubation using capnography

SECONDARY OUTCOMES:
The percentage of glottic opening (POGO) score | During anesthesia induction procedure
  The percentage of glottic opening (POGO), linear span from the anterior commissure to the interarytenoid notch, 0-100%
Cormack-Lehane grade | During anesthesia induction procedure
  The grade of glottic opening by intubation device (1= Full view of glottis, easy; 4=Neither glottis nor epiglottis seen, difficult)
Intubation difficulty scale (IDS) | During anesthesia induction procedure
  The intubation difficulty scale by the sum of seven variables (N1-N7). N1= the number of additional intubation attempts, N2= the number of additional operators, N3= the number of alternative intubation techniques used, N4= the laryngoscopic view, as defined by Cormack and Lehane, N5= the lifting force applied during laryngoscopy, N6= to the necessity to apply external laryngeal pressure to optimize glottic exposure, N7= vocal cord mobility. The IDS score is the sum of N1 through N7. The total IDS score ranges from zero (easy) to infinity (difficult).
Intubation difficulty by NRS score | During anesthesia induction procedure
  Intubation difficulty by NRS score (0=easy, 10=the most difficult)
Success rate in first attempt | During anesthesia induction procedure
  Successful intubation in a first attempt
Hemodynamic changes | During anesthesia induction procedure
  Blood pressure (mmHg) at 4 time points: Baseline, 1 minute after injection of anesthetic drugs, immediately before intubation, and 1 minute after intubation
Hemodynamic changes | During anesthesia induction procedure
  Heart rate (bpm) at 4 time points: Baseline, 1 minute after injection of anesthetic drugs, immediately before intubation, and 1 minute after intubation
Postoperative complications | An average of 1 hours after extubation
  Postoperative complications including sore throat, hoarseness/dysphonia, or pharyngeal pain

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Hospital, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No